CLINICAL TRIAL: NCT02369874
Title: A Phase III Randomized, Open-Label, Multi-Center, Global Study of MEDI4736 Monotherapy and MEDI4736 in Combination With Tremelimumab Versus Standard of Care Therapy in Patients With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: Study of MEDI4736 Monotherapy and in Combination With Tremelimumab Versus Standard of Care Therapy in Patients With Head and Neck Cancer
Acronym: EAGLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D4193C00002
Record Dates: First submitted 2015-02-18; First posted 2015-02-24 (Estimated); Results first posted 2019-10-03 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-01

CONDITIONS: Recurrent or Metastatic PD-L1-positive or -Negative Squamous Cell Carcinoma of the Head and Neck SCCHN
Keywords: Head and Neck cancer; MEDI4736; Tremelimumab
MeSH Terms: conditions — Recurrence; Head and Neck Neoplasms | interventions — durvalumab; tremelimumab; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MEDI4736 (Experimental): MEDI4736 monotherapy
  Interventions: Drug: MEDI4736
- MEDI4736 + Tremelimumab (Experimental): MEDI4736 + tremelimumab combination therapy
  Interventions: Drug: MEDI4736 + Tremelimumab
- Standard of Care (Active Comparator): Standard of Care
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: MEDI4736 — MEDI4736 Monotherapy
  Arms: MEDI4736
Drug: MEDI4736 + Tremelimumab — MEDI4736 + Tremelimumab combination therapy
  Arms: MEDI4736 + Tremelimumab
Drug: Standard of Care — Standard of Care
  Arms: Standard of Care

SUMMARY:
This is a randomized, open-label, multi-center, global, Phase III study to determine the efficacy and safety of MEDI4736 + tremelimumab combination therapy and MEDI4736 monotherapy versus SoC therapy in the target patient population.

DETAILED DESCRIPTION:
This is a randomized, open-label, multi-center, global, Phase III study to determine the efficacy and safety of MEDI4736 + tremelimumab combination therapy and MEDI4736 monotherapy versus SoC therapy in the target patient population.

The main objectives of the study are to:

* assess the efficacy of MEDI4736 + tremelimumab combination therapy versus SoC in patients with squamous cell carcinoma of the head and neck (SCCHN), in terms of overall survival (OS), regardless of PDL-1 status
* assess the efficacy of MEDI4736 monotherapy versus SOC in patients with SCCHN, in terms of OS, regardless of PDL-1 status

Patients will undergo a screening assessment on their tumor tissue sample to determine PD-L1 expression per a pre-specified cut-off level. Patients with ≥25% of tumor cells with membrane staining will be considered PD-L1 positive while those with 0% to 24% of tumor cells with membrane staining will be considered PD-L1 negative. Based on the underlying PD-L1 status, patients will be randomized in a 1:1:1 ratio to receive treatment with MEDI4736 monotherapy, MEDI4736 + tremelimumab combination therapy, or SoC therapy. Patients who discontinue treatment in 1 treatment group may not switch to treatment in a different group.

Stratification factors include PD-L1 status, human papillomavirus status, (in patients with oropharyngeal cancer only), and smoking status.

Tumor assessments will be performed every 8 weeks until objective tumor response by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1).

ELIGIBILITY:
Inclusion Criteria: - Age ≥18 years; - Written informed consent obtained from the patient/legal representative; - Histologically or cytologically confirmed recurrent or metastatic SCCHN; - Tumor progression or recurrence during or after only one palliative systemic treatment regimen for recurrent or metastatic disease that must have contained a platinum agent OR progression within 6 months of the last dose of platinum given as part of multimodality therapy with curative intent; - Confirmed PD-L1-positive or -negative SCCHN by the Ventana PD-L1 SP263 IHC assay; - WHO/Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1; At least 1 measurable lesion, - Not previously irradiated; - No prior exposure to immune-mediated therapy; - Adequate organ and marrow function; Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Exclusion Criteria: - Histologically or cytologically confirmed squamous cell carcinoma of any other primary anatomic location in the head and neck; - Received more than 1 palliative systemic regimen for recurrent or metastatic disease; -Any concurrent chemotherapy, Investigational Product, biologic, or hormonal therapy for cancer treatment; - Receipt of any investigational anticancer therapy within 28 days or 5 half-lives; - Receipt of last dose of an approved (marketed) anticancer therapy (chemotherapy, targeted therapy, biologic therapy, mAbs, etc) within 21 days prior to the first dose of study treatment; - Major surgical procedure within 28 days prior to the first dose of Investigational Product; - Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criterion; - Current or prior use of immunosuppressive medication within 14 days before the first dose of their assigned Investigational Product; - History of allogeneic organ transplantation; - Active or prior documented autoimmune or inflammatory disorders; - Uncontrolled intercurrent illness; - Patients with a history of brain metastases, spinal cord compression, or leptomeningeal carcinomatosis; - Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Fridericia's Correction; - History of active primary immunodeficiency; - Active tuberculosis; - Active infection including hepatitis B, hepatitis C or human immunodeficiency virus (HIV); - Receipt of live, attenuated vaccine within 30 days prior to the first dose of Investigational Product; - Pregnant or breast-feeding female patients; - Known allergy or hypersensitivity to Investigational Product

Ages: 18 Years to 96 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 736 (Actual)
Dates: Start 2015-09-09 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2020-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nassim Morsli, MD, Study Director — Medical Director AstraZeneca
Locations (147):
- United States (21):
  - Research Site, Tucson, Arizona
  - Research Site, Fullerton, California
  - Research Site, Los Angeles, California
  - Research Site, Redondo Beach, California
  - Research Site, Stanford, California
  - Research Site, Denver, Colorado
  - Research Site, Newark, Delaware
  - Research Site, Miami Beach, Florida
  - Research Site, Orlando, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Evanston, Illinois
  - Research Site, Lexington, Kentucky
  - Research Site, Boston, Massachusetts
  - Research Site, Rochester, New York
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Germantown, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, McAllen, Texas
  - Research Site, Norfolk, Virginia
- Argentina (2):
  - Research Site, CABA
  - Research Site, San Miguel de Tucumán
- Australia (5):
  - Research Site, Adelaide
  - Research Site, Heidelberg
  - Research Site, Melbourne
  - Research Site, St Leonards
  - Research Site, Woolloongabba
- Belgium (5):
  - Research Site, Brussels
  - Research Site, Charleroi
  - Research Site, Kortrijk
  - Research Site, Leuven
  - Research Site, Namur
- Brazil (7):
  - Research Site, Barretos
  - Research Site, Curitiba
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, Santo André
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Bulgaria (3):
  - Research Site, Shumen
  - Research Site, Sofia
  - Research Site, Varna
- Research Site, Temuco, Chile
- Croatia (2):
  - Research Site, Osijek
  - Research Site, Zagreb
- Czechia (2):
  - Research Site, Olomouc
  - Research Site, Zlín
- France (12):
  - Research Site, Angers
  - Research Site, Bordeaux
  - Research Site, Dijon
  - Research Site, Le Mans
  - Research Site, Lyon
  - Research Site, Montpellier
  - Research Site, Paris
  - Research Site, Plerin SUR MER
  - Research Site, Rouen
  - Research Site, Saint-Grégoire
  - Research Site, Strasbourg
  - Research Site, Villejuif
- Research Site, Lorient Cedex, Georgia
- Germany (8):
  - Research Site, Berlin
  - Research Site, Essen
  - Research Site, Halle
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Leipzig
  - Research Site, München
  - Research Site, Potsdam
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Győr
  - Research Site, Kecskemét
- Israel (5):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Petah Tikva
  - Research Site, Tel Aviv
  - Research Site, Tel Litwinsky
- Italy (9):
  - Research Site, Aosta
  - Research Site, Bologna
  - Research Site, Gallarate
  - Research Site, Legnago
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Pavia
  - Research Site, Roma
  - Research Site, Siena
- Japan (19):
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Hirakata-shi
  - Research Site, Isehara-shi
  - Research Site, Kashiwa
  - Research Site, Kitaadachi-gun
  - Research Site, Kobe
  - Research Site, Kōtoku
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Natori-shi
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Sapporo
  - Research Site, Sayama
  - Research Site, Shimotsuke-shi
  - Research Site, Sunto-gun
  - Research Site, Takatsuki-shi
  - Research Site, Yokohama
- Poland (3):
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Poznan
- Romania (4):
  - Research Site, Baia Mare
  - Research Site, Brasov
  - Research Site, Cluj-Napoca
  - Research Site, Craiova
- Russia (11):
  - Research Site, Arkhangelsk
  - Research Site, Chelyabinsk
  - Research Site, Kursk
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Omsk
  - Research Site, Pyatigorsk
  - Research Site, Saint Petersburg
  - Research Site, Sochi
  - Research Site, Ufa
  - Research Site, Vladimir
- Serbia (4):
  - Research Site, Belgrade
  - Research Site, Kamenitz
  - Research Site, Kragujevac
  - Research Site, Niš
- South Korea (4):
  - Research Site, Daegu
  - Research Site, Goyang-si
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (8):
  - Research Site, Barcelona
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Marbella
  - Research Site, Málaga
  - Research Site, Pamplona
  - Research Site, Valencia
  - Research Site, Zaragoza
- Taiwan (3):
  - Research Site, Kaohsiung City
  - Research Site, Taipei
  - Research Site, Taoynan
- Ukraine (5):
  - Research Site, Dnipro
  - Research Site, Kyiv
  - Research Site, Sumy
  - Research Site, Uzhhorod
  - Research Site, Zaporizhzhia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Ferris RL, Haddad R, Even C, Tahara M, Dvorkin M, Ciuleanu TE, Clement PM, Mesia R, Kutukova S, Zholudeva L, Daste A, Caballero-Daroqui J, Keam B, Vynnychenko I, Lafond C, Shetty J, Mann H, Fan J, Wildsmith S, Morsli N, Fayette J, Licitra L. Durvalumab with or without tremelimumab in patients with recurrent or metastatic head and neck squamous cell carcinoma: EAGLE, a randomized, open-label phase III study. Ann Oncol. 2020 Jul;31(7):942-950. doi: 10.1016/j.annonc.2020.04.001. Epub 2020 Apr 12. PMID 32294530
- See also: AstraZeneca Cancer Study Locator Service Phone: 877 400 4656 Email: astrazeneca@emergingmed.com — http://www.emergingmed.com/networks/AstraZeneca

RESULTS

PARTICIPANT FLOW:
Groups:
- Durvalumab + Tremelimumab: Participants received 20 mg/kg durvalumab and 1 mg/kg tremelimumab combination therapy via intravenous (IV) infusion every 4 weeks (q4w) for up to 16 weeks. 4 weeks after completion of combination therapy, participants received dosing with durvalumab 10 mg/kg monotherapy every 2 weeks (q2w) until disease progression (PD).
- Durvalumab: Participants received 10 mg/kg durvalumab via intravenous (IV) infusion every 2 weeks (q2w) until disease progression (PD).
- Standard of Care (SoC): Participants received monotherapy with 1 of the following therapies at the investigator's discretion until disease progression (PD): cetuximab, a taxane, methotrexate, or a fluoropyrimidine.
Period: Overall Study
Arm/Group | Durvalumab + Tremelimumab | Durvalumab | Standard of Care (SoC)
Started | 247 | 240 | 249
Received Treatment | 246 | 237 | 240
Completed | 203 | 183 | 188
Not Completed | 44 | 57 | 61
Not completed — Lost to Follow-up | 2 | 2 | 2
Not completed — Withdrawal by Subject | 7 | 9 | 27
Not completed — Miscellaneous | 1 | 1 | 0
Not completed — On Treatment/Off Study | 34 | 45 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Durvalumab + Tremelimumab | Durvalumab | Standard of Care (SoC) | Total
Number analyzed (Participants) | 247 | 240 | 249 | 736
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.9 (9.14) | 59.0 (10.07) | 59.5 (10.37) | 59.4 (9.86)
Age, Customized [Count of Participants; unit: Participants]
  < 65 Years | 174 | 169 | 171 | 514
  >= 65 - < 75 Years | 63 | 56 | 64 | 183
  >= 75 Years | 10 | 15 | 14 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 38 | 42 | 118
  Male | 209 | 202 | 207 | 618
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 15 | 13 | 44
  Not Hispanic or Latino | 226 | 223 | 229 | 678
  Unknown or Not Reported | 5 | 2 | 7 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 33 | 35 | 45 | 113
  Black Or African American | 1 | 0 | 3 | 4
  Other | 4 | 5 | 3 | 12
  White | 204 | 198 | 189 | 591
  Unknown or Not Reported | 5 | 2 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of randomization until death due to any cause. OS was analyzed for the full analysis set, regardless of programmed death-ligand 1 (PD-L1) status.
Time Frame: September 2015 to September 2018 (36 months)
Population: Full analysis set - inclusive of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab + Tremelimumab | Durvalumab | Standard of Care (SoC)
Number analyzed (Participants) | 247 | 240 | 249
Months | 6.5 [5.5 to 8.2] | 7.6 [6.1 to 9.8] | 8.3 [7.3 to 9.2]
Statistical Analysis 1: Comparison: Durvalumab + Tremelimumab vs Standard of Care (SoC); Test type: Superiority; p = 0.7624, Log Rank; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.85 to 1.26]
Statistical Analysis 2: Comparison: Durvalumab vs Standard of Care (SoC); Test type: Superiority; p = 0.1993, Log Rank; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.72 to 1.08]

2. Secondary Outcome: Overall Survival (OS) in PD-L1 Negative Participants
Description: OS is defined as the time from the date of randomization until death due to any cause. PD-L1 negative was defined as <25% of tumor cells with membrane staining for PD-L1 at any intensity.
Time Frame: September 2015 to September 2018 (36 months)
Population: PD-L1-negative analysis set - inclusive of all randomized participants whose PD-L1 status is PD-L1-negative as defined by the Ventana PD-L1 SP263 IHC assay.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab + Tremelimumab | Durvalumab | Standard of Care (SoC)
Number analyzed (Participants) | 175 | 172 | 177
Months | 7.8 [5.9 to 10.3] | 7.6 [6.2 to 9.5] | 8.0 [6.7 to 8.9]
Statistical Analysis 1: Comparison: Durvalumab + Tremelimumab vs Standard of Care (SoC); Test type: Superiority; p = 0.4590, Log Rank; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.73 to 1.17]
Statistical Analysis 2: Comparison: Durvalumab + Tremelimumab vs Durvalumab; Test type: Superiority; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.85 to 1.36]

3. Secondary Outcome: Overall Survival (OS) in PD-L1 Positive Participants
Description: OS is defined as the time from the date of randomization until death due to any cause. PD-L1 positive was defined as ≥25% of tumor cells with membrane staining for PD-L1 at any intensity.
Time Frame: September 2015 to September 2018 (36 months)
Population: PD-L1-positive analysis set - inclusive of all randomized participants whose PD-L1 status is PD-L1-positive as defined by the Ventana PD-L1 SP263 IHC assay.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab + Tremelimumab | Durvalumab | Standard of Care (SoC)
Number analyzed (Participants) | 72 | 68 | 72
Months | 4.8 [3.3 to 6.4] | 9.8 [4.3 to 14.1] | 9.0 [6.8 to 9.2]
Statistical Analysis 1: Comparison: Durvalumab vs Standard of Care (SoC); Test type: Superiority; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.63 to 1.39]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of randomization until the date of objective disease progression or death based on investigator assessments, according to response evaluation criteria in solid tumors 1.1 (RECIST1.1). Objective disease progression was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: September 2015 to September 2018 (36 months)
Population: Full analysis set - inclusive of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab + Tremelimumab | Durvalumab | Standard of Care (SoC)
Number analyzed (Participants) | 247 | 240 | 249
Months | 2.0 [1.9 to 2.3] | 2.1 [1.9 to 3.0] | 3.7 [3.1 to 3.7]
Statistical Analysis 1: Comparison: Durvalumab + Tremelimumab vs Standard of Care (SoC); Test type: Superiority; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.90 to 1.33]
Statistical Analysis 2: Comparison: Durvalumab vs Standard of Care (SoC); Test type: Superiority; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.84 to 1.25]

5. Secondary Outcome: Objective Response Rate (ORR)
Description: The percentage of participants who experienced an objective response (complete response [CR] or partial response [PR]), based on investigator assessments according to response evaluation criteria in solid tumors 1.1 (RECIST1.1). A CR was defined as the disappearance of all target lesions (TLs) since baseline. Any pathological lymph nodes selected as TLs must have a reduction in short axis to <10 mm. A PR was defined as at least a 30% decrease in the sum of the diameters of TLs, taking as reference the baseline sum of diameters.
Time Frame: Assessed at randomization and every 8 weeks thereafter
Population: Full analysis set - inclusive of all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Durvalumab + Tremelimumab | Durvalumab | Standard of Care (SoC)
Number analyzed (Participants) | 247 | 240 | 249
Percentage of participants | 18.2 [13.6 to 23.6] | 17.9 [13.3 to 23.4] | 17.3 [12.8 to 22.5]
Statistical Analysis 1: Comparison: Durvalumab + Tremelimumab vs Standard of Care (SoC); Test type: Superiority; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.67 to 1.70]
Statistical Analysis 2: Comparison: Durvalumab vs Standard of Care (SoC); Test type: Superiority; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.66 to 1.68]

6. Secondary Outcome: Duration of Response (DoR)
Description: Median DoR, in months, based on investigator assessments, according to response evaluation criteria in solid tumors 1.1 (RECIST1.1). A complete response was defined as the disappearance of all target lesions (TLs) since baseline. Any pathological lymph nodes selected as TLs must have a reduction in short axis to <10 mm. A partial response was defined as at least a 30% decrease in the sum of the diameters of TLs, taking as reference the baseline sum of diameters.
Time Frame: September 2015 to September 2018 (36 months)
Population: Full analysis set, participants with objective response - inclusive of all randomized participants with an objective response (RECIST 1.1).
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Durvalumab + Tremelimumab | Durvalumab | Standard of Care (SoC)
Number analyzed (Participants) | 45 | 43 | 43
Months | 7.4 [2.8 to NA] — Upper percentile not reached. | 12.9 [5.6 to NA] — Upper percentile not reached. | 3.7 [1.9 to 5.5]

7. Secondary Outcome: Disease Control Rate (DCR)
Description: 6 Months: The percentage of participants who had a best objective response of complete response (CR) or partial response (PR) in the first 6 months or had demonstrated stable disease (SD) for a minimum interval of 24 weeks following randomization.
  12 Months: The percentage of participants who had a best objective response of CR or PR within 12 months or had demonstrated SD for a minimum interval of 48 weeks following randomization.
  Objective response was based on investigator assessments, according to response evaluation criteria in solid tumors 1.1 (RECIST1.1). A CR was defined as the disappearance of all target lesions (TLs) since baseline. Any pathological lymph nodes selected as TLs must have a reduction in short axis to <10 mm. A PR was defined as at least a 30% decrease in the sum of the diameters of TLs, taking as reference the baseline sum of diameters.
Time Frame: Baseline up to 6 months; baseline up to 12 months
Population: Full analysis set - inclusive of all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Durvalumab + Tremelimumab | Durvalumab | Standard of Care (SoC)
Number analyzed (Participants) | 247 | 240 | 249
Percentage of participants
  6 Months | 25.1 | 24.2 | 24.9
  12 Months | 20.6 | 18.8 | 18.9
Statistical Analysis 1: Comparison: Durvalumab + Tremelimumab vs Standard of Care (SoC); 6 Month analysis; Test type: Superiority; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.67 to 1.52]
Statistical Analysis 2: Comparison: Durvalumab vs Standard of Care (SoC); 6 Month analysis; Test type: Superiority; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.64 to 1.46]
Statistical Analysis 3: Comparison: Durvalumab + Tremelimumab vs Standard of Care (SoC); 12 Month analysis; Test type: Superiority; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.72 to 1.75]
Statistical Analysis 4: Comparison: Durvalumab vs Standard of Care (SoC); 12 Month analysis; Test type: Superiority; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.63 to 1.57]

8. Secondary Outcome: Percentage of Participants Alive and Progression Free (APF)
Description: APF is defined as the percentage of participants who are alive and progression free at 6 months and 12 months after randomization. Estimates of progression free survival were based on investigator assessments according to response evaluation criteria in solid tumors 1.1 (RECIST1.1). Objective disease progression was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Baseline up to 6 months; baseline up to 12 months
Population: Full analysis set - inclusive of all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Durvalumab + Tremelimumab | Durvalumab | Standard of Care (SoC)
Number analyzed (Participants) | 247 | 240 | 249
Percentage of participants
  6 Months | 22.5 [17.4 to 28.0] | 25.1 [19.7 to 30.9] | 23.3 [17.8 to 29.3]
  12 Months | 11.0 [7.4 to 15.5] | 14.4 [10.1 to 19.5] | 5.7 [2.8 to 10.2]

9. Secondary Outcome: Percentage of Participants Alive
Description: Percentage of participants alive at 12, 18 and 24 months using a Kaplan Meier estimate.
Time Frame: 12, 18 and 24 months
Population: Full analysis set - inclusive of all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Durvalumab + Tremelimumab | Durvalumab | Standard of Care (SoC)
Number analyzed (Participants) | 247 | 240 | 249
Percentage of participants
  12 Months | 30.4 [24.7 to 36.3] | 37.0 [30.9 to 43.1] | 30.5 [24.7 to 36.4]
  18 Months | 21.0 [15.9 to 26.5] | 25.4 [19.9 to 31.3] | 17.8 [13.1 to 23.2]
  24 Months | 13.3 [8.9 to 18.6] | 18.4 [13.3 to 24.1] | 10.3 [5.7 to 16.5]

10. Secondary Outcome: Progression Free Survival (PFS) in PD-L1 Negative Participants
Description: Number of participants with confirmed objective disease progression (PD) at the time of the participant's last evaluable response evaluation criteria in solid tumors 1.1 (RECIST1.1) assessment. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. PD-L1 negative was defined as <25% of tumor cells with membrane staining for PD-L1 at any intensity.
Time Frame: September 2015 to September 2018 (36 months)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab + Tremelimumab | Durvalumab | Standard of Care (SoC)
Number analyzed (Participants) | 175 | 172 | 177
Participants | 154 | 151 | 144
Statistical Analysis 1: Comparison: Durvalumab + Tremelimumab vs Durvalumab; Test type: Superiority; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.76 to 1.21]

11. Secondary Outcome: Objective Response Rate (ORR) in PD-L1 Negative Participants
Description: The percentage of PD-L1 negative participants who experienced an objective response (complete response [CR] or partial response [PR]), based on investigator assessments according to response evaluation criteria in solid tumors 1.1 (RECIST1.1). A CR was defined as the disappearance of all target lesions (TLs) since baseline. Any pathological lymph nodes selected as TLs must have a reduction in short axis to <10 mm. A PR was defined as at least a 30% decrease in the sum of the diameters of TLs, taking as reference the baseline sum of diameters. PD-L1 negative was defined as <25% of tumor cells with membrane staining for PD-L1 at any intensity.
Time Frame: September 2015 to September 2018 (36 months)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Durvalumab + Tremelimumab | Durvalumab | Standard of Care (SoC)
Number analyzed (Participants) | 175 | 172 | 177
Percentage of participants | 17.7 [12.4 to 24.2] | 14.0 [9.1 to 20.0] | 15.3 [10.3 to 21.4]
Statistical Analysis 1: Comparison: Durvalumab + Tremelimumab vs Durvalumab; Test type: Superiority; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.74 to 2.39]

12. Secondary Outcome: Time to Deterioration in European Organisation for Research and Treatment of Cancer 30-item Core Quality of Life Questionnaire, Version 3 (EORTC QLQ-C30)
Description: The EORTC QLQ-C30 consists of 30 questions that can be combined to produce functional scales (e.g. physical), symptom scales (e.g. fatigue), and a global measure of health status. Each of the scales are measured from 0 to 100. Deterioration was defined as a 10-point decrease from baseline in a functioning or global health status/ quality of life score or a 10-point increase from baseline in a symptom score.
Time Frame: September 2015 to September 2018 (36 months)
Population: All randomized patients who provided questionnaire data
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab + Tremelimumab | Durvalumab | Standard of Care (SoC)
Number analyzed (Participants) | 227 | 226 | 227
Months
  Function - Physical: number analyzed (Participants) | 226 | 226 | 225
  Function - Physical | 2.0 [1.9 to 3.2] | 2.2 [1.9 to 3.5] | 3.7 [2.3 to 4.6]
  Symptom - Fatigue: number analyzed (Participants) | 220 | 220 | 218
  Symptom - Fatigue | 1.8 [1.3 to 1.9] | 1.4 [1.0 to 1.9] | 1.9 [1.6 to 2.6]
  Global health status/QoL: number analyzed (Participants) | 224 | 216 | 223
  Global health status/QoL | 1.9 [1.8 to 2.7] | 2.8 [1.9 to 3.8] | 3.5 [2.9 to 4.0]

13. Secondary Outcome: Time to Deterioration for European Organisation for Research and Treatment of Cancer 35-item Head and Neck Quality of Life Questionnaire (EORTC QLQ-H&N35)
Description: The EORTC QLQ-H&N35 comprises of 35 questions to assess head and neck cancer symptoms (e.g. pain, swallowing). Deterioration was defined as a 10-point increase from baseline in the symptom score.
Time Frame: September 2015 to September 2018 (36 months)
Population: All randomized patients who provided questionnaire data
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab + Tremelimumab | Durvalumab | Standard of Care (SoC)
Number analyzed (Participants) | 223 | 220 | 221
Months
  Pain (Mouth/ Throat): number analyzed (Participants) | 223 | 219 | 221
  Pain (Mouth/ Throat) | 2.9 [2.4 to 3.8] | 2.8 [2.6 to 3.7] | 3.4 [2.7 to 4.0]
  Swallowing: number analyzed (Participants) | 212 | 217 | 210
  Swallowing | 2.6 [1.9 to 3.6] | 2.8 [1.9 to 3.9] | 3.7 [2.9 to 4.6]

14. Secondary Outcome: Number of Participants Reporting One or More Adverse Events (AE)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. Inclusive of AEs and serious AEs.
Time Frame: First dose to last dose + 90 days or data cut off (up to 36 months)
Population: Safety analysis set - inclusive of all participants that received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab + Tremelimumab | Durvalumab | Standard of Care (SoC)
Number analyzed (Participants) | 246 | 237 | 240
Participants | 232 | 214 | 229

ADVERSE EVENTS:
Time Frame: First dose to last dose + 90 days or data cut off (maximum exposure 32 months)
Arm/Group | Durvalumab + Tremelimumab | Durvalumab | Standard of Care (SoC)
All-Cause Mortality (participants affected / at risk) | 206/247 | 186/240 | 199/249
Serious Adverse Events (participants affected / at risk) | 79/246 | 69/237 | 61/240
Other Adverse Events (participants affected / at risk) | 203/246 | 180/237 | 207/240
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab + Tremelimumab (N=246) | Durvalumab (N=237) | Standard of Care (SoC) (N=240)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 2 (2) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophageal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Stoma site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Abdominal wall wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Osteoradionecrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Acquired tracheo-oesophageal fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Coeliac disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1)
Gastric fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Tongue haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (1) | 1 (1)
Chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Death (General disorders) | 2 (2) | 2 (2) | 2 (2)
Facial pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 4 (4) | 1 (1)
Hyperthermia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 2 (2) | 2 (2)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abscess oral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (3)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 2 (2) | 2 (2)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 9 (9) | 8 (9) | 9 (9)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 4 (4) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 0 (0) | 4 (4)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Streptococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Nasal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Petroleum distillate poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 2 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (5) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 4 (4) | 2 (2)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Carotid artery disease (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Horner's syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 1 (1)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Hallucinations, mixed (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 3 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (6) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 3 (3)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Vasculitic ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 2 (2) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab + Tremelimumab (N=246) | Durvalumab (N=237) | Standard of Care (SoC) (N=240)
Anaemia (Blood and lymphatic system disorders) | 55 (68) | 47 (57) | 56 (94)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3) | 8 (10) | 20 (25)
Leukopenia (Blood and lymphatic system disorders) | 10 (19) | 2 (3) | 13 (42)
Neutropenia (Blood and lymphatic system disorders) | 11 (16) | 4 (4) | 32 (86)
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (23) | 5 (11) | 18 (49)
Hypothyroidism (Endocrine disorders) | 32 (33) | 33 (44) | 5 (5)
Constipation (Gastrointestinal disorders) | 33 (37) | 33 (40) | 29 (29)
Diarrhoea (Gastrointestinal disorders) | 38 (50) | 24 (46) | 32 (42)
Dysphagia (Gastrointestinal disorders) | 20 (22) | 28 (30) | 18 (18)
Nausea (Gastrointestinal disorders) | 30 (36) | 27 (29) | 41 (47)
Stomatitis (Gastrointestinal disorders) | 5 (7) | 11 (12) | 27 (34)
Vomiting (Gastrointestinal disorders) | 15 (16) | 18 (23) | 20 (24)
Asthenia (General disorders) | 51 (57) | 42 (53) | 56 (63)
Fatigue (General disorders) | 40 (44) | 31 (35) | 35 (44)
Mucosal inflammation (General disorders) | 2 (3) | 3 (3) | 17 (20)
Pyrexia (General disorders) | 31 (35) | 19 (23) | 29 (42)
Alanine aminotransferase increased (Investigations) | 15 (20) | 11 (11) | 17 (28)
Aspartate aminotransferase increased (Investigations) | 15 (17) | 7 (8) | 14 (23)
Blood alkaline phosphatase increased (Investigations) | 14 (20) | 7 (11) | 8 (9)
Gamma-glutamyltransferase increased (Investigations) | 17 (18) | 9 (11) | 12 (19)
Weight decreased (Investigations) | 27 (27) | 31 (33) | 20 (22)
Decreased appetite (Metabolism and nutrition disorders) | 44 (51) | 30 (33) | 48 (56)
Hypercalcaemia (Metabolism and nutrition disorders) | 17 (21) | 10 (12) | 7 (8)
Hyponatraemia (Metabolism and nutrition disorders) | 14 (16) | 11 (15) | 8 (8)
Neck pain (Musculoskeletal and connective tissue disorders) | 20 (20) | 15 (16) | 23 (24)
Headache (Nervous system disorders) | 11 (11) | 13 (15) | 16 (19)
Neuropathy peripheral (Nervous system disorders) | 4 (4) | 5 (5) | 24 (26)
Insomnia (Psychiatric disorders) | 13 (13) | 7 (7) | 8 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 26 (27) | 25 (26) | 19 (22)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 27 (27) | 27 (29) | 19 (21)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 29 (30)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 17 (18)
Pruritus (Skin and subcutaneous tissue disorders) | 23 (28) | 10 (13) | 9 (10)
Rash (Skin and subcutaneous tissue disorders) | 18 (20) | 19 (22) | 36 (38)
Hypertension (Vascular disorders) | 17 (17) | 11 (14) | 7 (8)

LIMITATIONS AND CAVEATS:
Multiple testing was performed for OS analysis in the intent-to-treat (ITT) population and OS analysis in the PD-L1 negative population for durvalumab + tremelimumab versus SoC only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-01-18): https://cdn.clinicaltrials.gov/large-docs/74/NCT02369874/SAP_000.pdf
  • Study Protocol (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/74/NCT02369874/Prot_001.pdf